CLINICAL TRIAL: NCT06273293
Title: Postprocedural Contrast Mediated FFR Plus Intracoronary Infusion of Nitroglycerin in Multivessel Patients
Brief Title: Postprocedural Contrast Mediated FFR Plus Intracoronary Infusion of Nitroglycerin in Multivessel Patients (PROMETEUS TRIAL)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fundación EPIC (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: EPIC35-PROMETEUS
Record Dates: First submitted 2024-02-15; First posted 2024-02-22 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Coronary Disease
Keywords: Percutaneous Coronary Intervention (PCI); Fractional Flow Reserve
MeSH Terms: conditions — Coronary Disease | interventions — Fractional Flow Reserve, Myocardial

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Percutaneous coronary intervention (PCI) and guide wire post PCI in multivessel patients (Other)
  Interventions: Diagnostic Test: Fractional Flow Reserve

INTERVENTIONS:
Diagnostic Test: Fractional Flow Reserve — Agreement measurements between the different post-ICP functional values (cFFR+NTG and FFR) will be performed at the end of the intervention on the treated vessels. The study protocol consists of 4 sequential steps (separated by at least 30 sec):
  1. Determination of FFR with contrast and NTG: cFFR +NTG will be calculated with the lowest ratio after the infusion of 0.2 mg bolus of intracoronary NTG and pushed with contrast.
  2. Determination of distal pressure between basal aortic pressure: The Pd/Pa will be obtained after about 30-60 seconds of the NTG bolus in step 1.
  3. Determination of the diastolic dPR index: the average value (2-3 determinations).
  4. Determination of fractional flow reserve with adenosine: The FFR will be obtained after continuous peripheral venous infusion with adenosine or with intracoronary boluses according to the protocol of each center.

SUMMARY:
the use of pressure wires is the standar of care to evaluate angiographically intermediate coronary lesions, however, limitations in the management of these type of lesions continue to be a challenge for the interventional cardiologist. The use of FFR has some limitations such as the use of adenosine due to its cost, adverse effects (e.g. transient atrioventricular block, angina, headache, etc.), time consuming and some relative contraindications for its use. In this sense, in recent years new rest indices (iFR, RFR, dPR) and hyperemic indices without adenosine (cFFR-NTG, Pd/Pa-NTG or cFFR) have been developed, demonstrating an improvement in terms of outcomes with its use, so they can also be used as a tool to guide us to plan our strategy. These new indices, particularly the cFFR-NTG, are simpler, at least as safe and have an excellent correlation with the FFR with adenosine in the assessment of intermediate coronary lesions.

In recent years, functional assessment after intervention has also been increasingly implemented, which, like intracoronary imaging, can make us change our attitude and correlate with the prognosis. The lower implementation of this practice, especially in multivessel patients, may result from having to lose the position of the wire to check equalization, difficulty in crossing the wire, wear/breakage of the material after diagnosis (2-3 vessels), use more time and contrast, etc. These problems could be reduced, at least partially, with the use of the workhorse coronary guidewire pressure microcatheter to measure post-PCI functional assessment. Although the usefulness of post-PCI FFR has been demonstrated, there is no clearly established cut-off value (0.84-0.96) and it seems that in reality the values are a continuum of risk so that the higher the value, the better the prognosis . Furthermore, other simpler indices such as rest or hyperemic indices without adenosine have not been correlated with FFR in post-PCI.

The purpose of this study is to evaluate the correlation between cFFR-NTG and other indices taking FFR as a reference in multivessel patients after undergoing intervention. Establish cut-off points and correlate it with adverse cardiovascular events (MACE) in a 1-year clinical follow-up.

DETAILED DESCRIPTION:
Percutaneous coronary intervention (PCI) is a standard treatment strategy for coronary artery disease (CAD). With the presence of myocardial ischemia, PCI reduces the risks of death, myocardial infarction (MI), and revascularization compared to medical therapy. However, the risk of future clinical events remains high, and about 10% of patients experienced further cardiovascular events after PCI. Facing intermediate coronary lesions the use of pressure wires is the standar of care, however, limitations in the management of angiographically intermediate coronary lesions continue to be a challenge for the interventional cardiologist. The measurement of fractional flow reserve (FFR) to determine the hemodynamic relevance of coronary stenosis has been shown to be a technique that improves the prognosis and cost-efficiency of the procedures when compared to visual angiographic interpretation alone. Due to this evidence, the use of FFR to guide interventional procedures is a class I recommendation in current clinical practice guidelines.

Patients with multivessel coronary artery disease are another field in the use of pressure guiding. In these patients, the use of FFR has demonstrated the reclassification of the severity of coronary lesions in up to 40% of cases, modifying the number of functionally significant lesions and making it possible to reorient therapeutic decisions, avoiding interventional treatment of non-significant lesions and with a better prognosis.

However, the use of FFR has some limitations such as the use of adenosine due to its cost, adverse effects (e.g. transient atrioventricular block, angina, headache, etc.) and time consuming. In addition, the presence of atrioventricular block, asthma or severe chronic obstructive pulmonary disease are relative contraindications for its use. In this sense, in recent years new rest indices (iFR, RFR, dPR) and hyperemic indices without adenosine (cFFR-NTG, Pd/Pa-NTG or cFFR) have been developed , demonstrating an improvement in terms of outcomes with its use, so they can also be used as a tool to guide us to plan our strategy. These new indices, particularly the cFFR-NTG, are simpler, at least as safe and have an excellent correlation with the FFR with adenosine in the assessment of intermediate coronary lesions.

In recent years, functional assessment after intervention has also been increasingly implemented, which, like intracoronary imaging, can make us change our attitude and correlate with the prognosis. The lower implementation of this practice, especially in multivessel patients, may result from having to lose the position of the wire to check equalization, difficulty in crossing the wire, wear/breakage of the material after diagnosis (2-3 vessels), use more time and contrast, etc. These problems could be reduced, at least partially, with the use of the workhorse coronary guidewire pressure microcatheter to measure post-PCI functional assessment. Although the usefulness of post-PCI FFR has been demonstrated, there is no clearly established cut-off value (0.84-0.96) and it seems that in reality the values are a continuum of risk so that the higher the value, the better the prognosis . Furthermore, other simpler indices such as rest or hyperemic indices without adenosine have not been correlated with FFR in post-PCI.

The purpose of this study is to evaluate the correlation between cFFR-NTG and other indices taking FFR as a reference in multivessel patients after undergoing intervention. Establish cut-off points and correlate it with adverse cardiovascular events (MACE) in a 1-year clinical follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Patients >18 years old and,
* Patients with multivessel coronary artery disease (multivessel coronary artery disease will be considered the presence of significant stenosis in 2 or more first or second order vessels greater than 1.5 mm in diameter with an angiographic reduction of their diameter ≥50% by visual estimation) subsidiary of percutaneous coronary revascularization in at least one of them and,
* Use of Navvus pressure microcatheter both for functional diagnosis and for post-PCI evaluation of the different vessels and,
* Patients who have signed the Informed Consent.

Exclusion Criteria:

* Patients with intolerance or contraindication to adenosine.
* Hemodynamically unstable patients, acute phase of a STEACS.
* Patient with significant comorbidity with limited life expectancy.
* Patients with the patient's express refusal to participate in the study.
* Pregnant or breastfeeding female patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-05-31 (Actual); Primary Completion 2025-12-20 (Estimated); Study Completion 2026-01-20 (Estimated)

PRIMARY OUTCOMES:
Agreement between cFFR+NTG and FFR | Index Procedure
  To evaluate the agreement between cFFR+NTG and FFR after successful angiographic revascularization of lesions in multivessel patients.
SAFETY: MACE | 12 months
  To evaluate the safety associated with performing PCI in multivessel patients with a pre- and post-PCI functional study in terms of MACE at 12 months that includes: Cardiovascular death, Acute myocardial infarction of the lesion treated/functionally evaluated, Need for revascularization of the treated/functionally evaluated lesion.

SECONDARY OUTCOMES:
Agreement between Pd/Pa or dPR and FFR | Index Procedure
  To evaluate the agreement between Pd/Pa or dPR and FFR after successful angiographic revascularization of lesions in multivessel patients, with a cut-off point of FFR ≥0.80.
Cut-off point for cFFR+NTG post-ICP | Index Procedure
  Determine a cut-off point for cFFR+NTG post-ICP.
Evaluate the change in strategy that the measurement of FFR values ≤0.90 post-PCI | Index Procedure
  Evaluate the change in strategy that the measurement of FFR values ≤0.90 post-PCI may entail: use of intracoronary imaging techniques, post-dilation, etc.
Cardiac death | 12 months
  Cardiac death
Cardiovascular death | 12 months
  Cardiovascular death
Acute myocardial infarction of the lesion treated/functionally evaluated | 12 months
  Acute myocardial infarction of the lesion treated/functionally evaluated
Acute myocardial infarction from any lesion | 12 months
  Acute myocardial infarction from any lesion
Need for revascularization of the lesion treated/functionally evaluated | 12 months
  Need for revascularization of the lesion treated/functionally evaluated
Need for revascularization of any lesion | 12 months
  Need for revascularization of any lesion

CONTACTS AND LOCATIONS:
Locations (4):
- Spain (4):
  - Hospital Universitario San Juan de Alicante, Alicante
  - Hospital Universitario de Badajoz, Badajoz
  - Hospital Universitario Juan Ramón Jiménez, Huelva
  - Hospital Universitario Virgen del Rocío, Seville

REFERENCES:
- [Background] Neumann FJ, Sousa-Uva M, Ahlsson A, Alfonso F, Banning AP, Benedetto U, Byrne RA, Collet JP, Falk V, Head SJ, Juni P, Kastrati A, Koller A, Kristensen SD, Niebauer J, Richter DJ, Seferovic PM, Sibbing D, Stefanini GG, Windecker S, Yadav R, Zembala MO; ESC Scientific Document Group. 2018 ESC/EACTS Guidelines on myocardial revascularization. Eur Heart J. 2019 Jan 7;40(2):87-165. doi: 10.1093/eurheartj/ehy394. No abstract available. PMID 30165437
- [Background] van Nunen LX, Zimmermann FM, Tonino PA, Barbato E, Baumbach A, Engstrom T, Klauss V, MacCarthy PA, Manoharan G, Oldroyd KG, Ver Lee PN, Van't Veer M, Fearon WF, De Bruyne B, Pijls NH; FAME Study Investigators. Fractional flow reserve versus angiography for guidance of PCI in patients with multivessel coronary artery disease (FAME): 5-year follow-up of a randomised controlled trial. Lancet. 2015 Nov 7;386(10006):1853-60. doi: 10.1016/S0140-6736(15)00057-4. Epub 2015 Aug 30. PMID 26333474
- [Background] Gutierrez-Barrios A, Noval-Morillas I, Camacho-Freire S, Puche JE, Gheorghe L, Silva E, Alarcon-Lastra I, Canadas-Pruano D, Gomez-Menchero A, Calle-Perez G, Diaz-Fernandez JF, Vazquez-Garcia R. Contrast FFR plus intracoronary injection of nitro-glycerine accurately predicts FFR for coronary stenosis functional assessment. Minerva Cardiol Angiol. 2021 Aug;69(4):449-457. doi: 10.23736/S2724-5683.20.05354-2. Epub 2020 Dec 1. PMID 33258564
- [Background] Patel MR, Jeremias A, Maehara A, Matsumura M, Zhang Z, Schneider J, Tang K, Talwar S, Marques K, Shammas NW, Gruberg L, Seto A, Samady H, Sharp ASP, Ali ZA, Mintz G, Davies J, Stone GW. 1-Year Outcomes of Blinded Physiological Assessment of Residual Ischemia After Successful PCI: DEFINE PCI Trial. JACC Cardiovasc Interv. 2022 Jan 10;15(1):52-61. doi: 10.1016/j.jcin.2021.09.042. PMID 34991824
- [Background] Thakur U, Khav N, Comella A, Michail M, Ihdayhid AR, Poon E, Nicholls SJ, Ko B, Brown AJ. Fractional Flow Reserve following Percutaneous Coronary Intervention. J Interv Cardiol. 2020 Jun 5;2020:7467943. doi: 10.1155/2020/7467943. eCollection 2020. PMID 32565755